CLINICAL TRIAL: NCT06881303
Title: Impact of Prior Identification and Education of Patients Requiring a Digestive Stoma for Fecal Diversion
Acronym: RESTODIG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RCAPHM23_0029; 2023-A01631-44 (Other: IDRCB)
Record Dates: First submitted 2025-03-05; First posted 2025-03-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Anastomosis; Endometrial; Anastomotic Leak Rectum; Ulcerative Colitis (Disorder); Adenomatous Polyposis Coli, Familial; Crohn Disease; Digestive Cancers; Protectomy
MeSH Terms: conditions — Colitis, Ulcerative; Adenomatous Polyposis Coli; Crohn Disease; Gastrointestinal Neoplasms | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative identification and education (Experimental)
  Interventions: Other: preoperative stoma identification and education
- lack of preoperative identification and education (No Intervention)

INTERVENTIONS:
Other: preoperative stoma identification and education — The guide to good stoma therapy practice recommends that the site of the future stoma should be marked out preoperatively, in the lying, sitting and standing positions, so that the patient can see the stoma. What's more, the psychological impact of the stoma is such that preoperative and regular postoperative education is essential. This identification and initiation of education is carried out by stoma nurses and/or surgeons.
  Arms: Preoperative identification and education

SUMMARY:
There are many indications for performing a fecal diversion stoma. In both scheduled and emergency situations, and whatever the context (indication or type of fecal diversion stoma), stomal complications can occur early (10-60%) or late (25%), and may require repeat surgery. The most frequent complications are necrosis, retraction, bleeding, evisceration, occlusion, abscess, hyperflow with hydroelectrolytic consequences, skin lesions, prolapse or eventration. What's more, a temporary stoma can become permanent.

The positioning and fabrication of the digestive stoma for fecal diversion must therefore comply with well-defined criteria to reduce the risk of stomal complications and the difficulties of fitting the stoma, and thus improve the autonomy and therefore the quality of life of the ostomate patient. The guide to good stoma therapy practice recommends that the site of the future stoma should be marked out preoperatively. What's more, the psychological impact of a stoma is such that preoperative and regular postoperative education is essential. This identification and initiation of education is carried out by stoma nurses and/or surgeons.

The impact of preoperative stoma identification and education on stoma complications, quality of life and patient autonomy has been reported in a few comparative series. The impact of preoperative education on quality of life has also been reported.

However, despite this "Evidence Based Medicine", and the guide to good stoma therapy practice, the identification and education of the future fecal diversion stoma are not always carried out preoperatively. Reasons for this may include lack of time, lack of human resources, in the general context of a shrinking public hospital, or in the current context of distancing and dehumanization of the profession, or lack of conviction on the part of practitioners.

To this end, the investigators would like to propose a prospective observational study aimed at evaluating the impact of identification and education prior to the performance of a fecal diversion stoma in a programmed situation on the one hand, and an emergency situation on the other.

The main objective will be to compare quality of life specifically related to the stoma at 30 days postoperatively with the StomaQOL score, between 2 groups of patients:

* unexposed group: no preoperative stoma identification and education
* exposed group: preoperative stoma identification and education. This comparison will be stratified according to whether surgery is scheduled or emergency surgery.

Total 100 patients :

* In scheduled surgery: 30 exposed and 30 unexposed patients
* In emergency surgery: 10 exposed and 30 unexposed patients

Timeline:

Inclusion period: 12 months Follow-up period: 12 months Total duration: 24 months

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 and over
* for whom a fecal diversion stoma is planned on a scheduled or emergency basis
* affiliated with the French social security system

Exclusion Criteria:

* Patient in a period of exclusion from another research protocol at the time of signing the no-objection form,
* Subjects covered by articles L1121-5 to 1121-8 of the French Public Health Code (minors, adults under guardianship or trusteeship, patients deprived of their liberty, pregnant or breast-feeding women),
* No digestive stoma or fecal diversion planned
* Person who does not understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Questionnary : quality of life | From enrollment to the end of the study at 24 months

SECONDARY OUTCOMES:
occurrence of short-term stomatal complications (within 30 days days post-operatively) | From intervention to 30 days after intervention
  edema, necrosis, retraction, bleeding, evisceration, occlusion, abscess, hyperflow with hydroelectrolytic consequences, skin lesions
Questionnaire about the patient's autonomy when returning home (stoma therapist needed or not; if present, for how long) | From intervention to 30 days after intervention
  stoma therapist needed or not; if present, for how long
rate of long-term stomatal complications at 1 year | From intervention to1 year after intervention
  prolapse, occlusion, ventration
questionnaire on ostomy-specific quality of life, assessed by the StomaQOL score at 30 days, for comparison between identification and education by the stoma nurse or surgeon | From intervention to 30 days after intervention
Questionnaire on ostomy-specific quality of life, assessed by the StomaQOL score at 1 years | From intervention to 1 year after intervention
SF36 quality of life questionnaire at 30 days and 1 year | From intervention to 1 year after intervention
Rate of restoration of digestive continuity at 1 year | From intervention to 1 year after intervention
Reasons for not carrying out preoperative identification and education | From enrollment to the end of the study at 24 months
  emergency, surgery at night or on weekends or public holidays, insufficient preoperative time, stoma nurse absent, surgeon's choice, patient's wishes.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance publique - Hôpitaux de Marseille, Marseille, France